CLINICAL TRIAL: NCT00925808
Title: A Prospective Study of Cancer Patients Diagnosed With Unsuspected Venous Thromboembolism (VTE) on Routine Computed Tomography (CT) Scans
Brief Title: Cancer Patients Diagnosed With Unsuspected Venous Thromboembolism (VTE) on Routine Computed Tomography (CT) Scans
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0026
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Cancer; Venous Thromboembolism
Keywords: Unsuspected Venous Thromboembolism; VTE; Routine Computed Tomography; CT Scans
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unsuspected VTE: Prevalence of unsuspected VTE in oncology patients on routine staging CT scans of the thorax, abdomen and pelvis
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Survey tools and VTE Symptom Follow-up Questionnaire

SUMMARY:
This is a prospective study with the following objectives:

Primary Objective:

1. To estimate the prevalence of unsuspected VTE in oncology patients on routine staging CT scans of the thorax, abdomen and pelvis.

   Secondary Objectives:
2. To identify symptoms commonly associated with VTE that are present in cancer patients undergoing routine staging CT scans with findings of unsuspected VTE.
3. To identify the risk factors and demographic characteristics in outpatient cancer patients associated with the development of unsuspected VTE.
4. To determine the incidence of recurrence of new VTE in patients with unsuspected VTE at 3 and 6 months of follow-up.

DETAILED DESCRIPTION:
Patients diagnosed with cancer are routinely scheduled for staging CT scans. The CT scans are obtained to stage a new cancer diagnosis, to restage a cancer after treatment initiation or to evaluate abnormal masses, disease progression or metastasis. The study population will include outpatients scheduled for routine CT scan of the chest, abdomen and/or pelvis.

While patients are waiting in the Diagnostic Imaging waiting area, they will be invited to participate in the study. Study eligibility will be determined by administering a screening questionnaire. Cancer patients who meet the eligibility criteria will be asked to participate in the study. It is imperative that the patient completes the surveys and not the caregiver. A caregiver may lend assistance in transcribing the information but may not complete the instruments independent of the patient.

Many of these tools are brief and the estimated completion time should be approximately 15 to 30 minutes. Additionally completing the instruments will not extend beyond the time the patient is in the CT scan waiting area prior to the scheduled study.

On the day of study enrollment, patients will be asked to complete Brief Fatigue Inventory (BFI), MD Anderson Symptom Inventory (MDASI), Dyspnea Numerical Scale (DNS), Cancer Dyspnea Scale (CDS), ECOG/Zubrod Performance scale, Depression Anxiety Stress Scale (DASS 21), VTE Symptom Enrollment Questionnaire and Functional Assessment of Cancer Therapy-General (FACT-G). The patients will also complete a questionnaire on symptoms of VTE such as chest pain, pain or swelling of the extremities and other common symptoms reported in VTE patients.

VTE Symptom Follow-up Questionnaire:This instrument was designed for this study. Patients will be asked at 3 and 6 months the treatments received, recurrence of VTE, incidence of bleeding episodes and other health related conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of cancer.
2. Subjects must be 18 years or more.
3. Male and female patients are eligible for enrollment.
4. Patients who are scheduled for routine outpatient cancer staging using CT scans.
5. Patients must be able to complete the required survey tools independently.
6. Patients must be able to speak, read and write English.

Exclusion Criteria:

1. Patients who have a clinically suspected VTE and/or scheduled for CT scans for suspected VTE.
2. Patients not willing to complete survey tools.
3. Prior history of PE or DVT.
4. Eastern Cooperative Oncology Group (ECOG)/Zubrod Performance Status score of 4.
5. Patients currently on anticoagulation therapy (low molecular weight heparin, fondaparinux, dalteparin, warfarin or unfractionated heparin). Patients on heparin flushes for indwelling catheters will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include cancer outpatients, 18 years or older, scheduled for routine CT scan of the chest, abdomen and/or pelvis at UT MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 1187 (Estimated)
Dates: Start 2009-06 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Unsuspected Venous Thromboembolism (VTE) Rate | Day of enrollment, 3 months (+/- 7 days) and 6 months (+/- 7 days) from study enrollment and during 3 and 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Escalante, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org